CLINICAL TRIAL: NCT06958068
Title: Integrating Mandatory Sexual Health Counseling in Gynaecological Oncology: A Paradigm Shift From Diagnosis to Survivorship.
Brief Title: Sexual Health Integration in Treatment of Gynecological Oncology
Acronym: SHIFT-GO
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Krzysztof Nowosielski, profesor, Medical University of Silesia
Other Study IDs: KB/96/FI/2018
Record Dates: First submitted 2025-04-27; First posted 2025-05-06 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Cervical Cancers; Vaginal Cancers; Sexual Health Quality of Life; Sexual Counselling
Keywords: gynecological cancer; sexual health; sexual counselling; paradigma; sexual activity
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Vaginal Neoplasms; Sexual Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women diagnosed with gynecological cancer after treatment completion: Observational questionnaire-based study

SUMMARY:
The goal of this cross-section observational and questionary based study is to learn how geological cancer survivors perceive sexual health support given by health care professionals during diagnosis and treatment process.

The main question to be answered is:

Who, when and to what extend should discuss the sexual health issues

The participants will answer online survey questions about Sexual health issues and Sexual counselling during diagnosis, treatment and follow-up.

DETAILED DESCRIPTION:
The main aim of the study is to verify who, from medical specialist, should discuss the sexual health issues in gynecological cancer survivors, when that discussion should take places and to what exited all sexual issues should be discusses.

The secondary end points are:

* to establish factors affecting returning to sexual activities defined as any type of physical contact with a partner engaging sexual organs as well as mutual and solo masturbation.
* to verified if gender of counselling specialist is important to patients.

The study is a cross-section observation one. It is based on a survey containing questions regarding basic socioeconomical factors, treatment history, reproductive history, and those concerning the opinion who, when, to what extend and how should ask about sexual issues during therapy modalities planning, treatment and follow-up.

Women after completing a treatment irrespectively of its type (surgery, radiation, chemotherapy, immune check point inhibitors) will be eligible for the study. Those who are no more sexually active and currently have no sexual partner will also be included.

After collecting the date three main analysis will be conducted to answer the study questions.

The results will be used as a basic for further work on recommendation on sexual health counselling in gynecological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with gynecological malignancies except breast cancer
* completion of treatment irrespectively of its type (surgery, CTH, RTH, immunotherapy)
* ECOG≤2

Exclusion Criteria:

* diagnosed with breast cancer
* currently being treated for gynecological or other malignancies
* ECOG >2
* not being able to have any type of sexual activity due to physical limitations or comorbidities

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with ovarian, cervical, endometrial, vulvar and vaginal cancer after completion of treatment irrespectively of its type (surgery, CTH, RTH, immunotherapy)
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Who should counsel patients with gynecological malignancies | At least 8 weeks post treatment completion
  A set of questions were asked to verify the hypothesis that specialist in gynecological oncology should inform about sexual issues during the treatment ant after its completion. Timing, frequency of counselling and patients' preferences for sexual information sources were established.

SECONDARY OUTCOMES:
Gender of gynecological oncologist counselling the patient | At least 8 weeks post treatment completion
  A set of questions were ask to verify the hypothesis that in case of cancer choosing the specialist in gynecological oncology in not gender-based but knowledge and skills-based.
Returning to sexual activity defining as any sexual contact with a partner or solo masturbation | At least 8 weeks post treatment completion
  A set of question were asked to verify factors that might influence returning to sexual activity after treatment completion

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynaecology, Obstetrics and Gynaecological Oncology, University Clinical Centre, Medical University of Silesia, Katowice, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
All anonymized data will be available
Supporting Information: Study Protocol, CSR
Time Frame: 31.12.2025
Access Criteria: On request

REFERENCES:
- [Background] Kowalczyk R, Nowosielski K, Cedrych I, Krzystanek M, Glogowska I, Streb J, Kucharz J, Lew-Starowicz Z. Factors Affecting Sexual Function and Body Image of Early-Stage Breast Cancer Survivors in Poland: A Short-Term Observation. Clin Breast Cancer. 2019 Feb;19(1):e30-e39. doi: 10.1016/j.clbc.2018.09.006. Epub 2018 Sep 21. PMID 30385228
- [Background] Kacperczyk-Bartnik J, Nowosielski K, Razumova Z, Bizzarri N, Pletnev A, Lindquist D, Lanner M, Nikolova T, Theofanakis C, Strojna AN, Bartnik P, Gomez-Hidalgo NR, Vlachos DE, Selcuk I, Zalewski K. Clinician attitude towards sexual counseling in women with gynecologic malignancies: European Network of Young Gynaecological Oncologists (ENYGO) survey. Int J Gynecol Cancer. 2022 Oct 3;32(10):1309-1315. doi: 10.1136/ijgc-2021-003309. PMID 35568382
- [Background] Nowosielski K, Palka A. Couples' sexual health after gynaecological cancer diagnosis - an unexplored area for further research. Contemp Oncol (Pozn). 2023;27(1):47-56. doi: 10.5114/wo.2023.127308. Epub 2023 Apr 27. PMID 37266338